CLINICAL TRIAL: NCT02044562
Title: Study of Dietary Nitrate on Plasma Nitrate Levels for Nasopharyngeal Carcinoma Patients Receiving Concurrent Chemo-radiotherapy
Brief Title: Dietary Nitrate on Plasma Nitrate Levels for Nasopharyngeal Carcinoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Songlin Wang, Professor and Vice President, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-07-08
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: dietary nitrate; radiotherapy; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nitrate supplementation (Experimental): Patients will receive 7-day nitrate supplementation at the end of the radiotherapy.
  Interventions: Dietary Supplement: nitrate supplementation
- Placebo (Placebo Comparator): Patients will receive 7-day placebo supplementation at the end of the radiotherapy
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: nitrate supplementation — A 70 ml beetroot juice containing 0.45g nitrate will be provided to the patients for 7 days at the end of the radiotherapy.
  Arms: nitrate supplementation
Dietary Supplement: Placebo — A 70 ml placebo containing 0 g nitrate will be provided to the patients for 7 days at the end of the radiotherapy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether dietary nitrate supplementation could improve the plasma nitrate levels for nasopharyngeal carcinoma patients receiving concurrent chemo-radiation therapy.

DETAILED DESCRIPTION:
Twenty patients diagnosed as nasopharyngeal carcinoma will be recruited. A 70 ml beetroot juice containing 0.45g nitrate or placebo will be provided to the patients for 7 days at the end of the radiotherapy . The plasma nitrate levels will be determined before radiotherapy, before intervention and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stages III-IVb (UICC 2002) nasopharyngeal carcinomas, will be recruited.

Exclusion Criteria:

* Patients with local invasion or metastatic foci in salivary glands, detected by MRI and PET-CT prior to treatment, were excluded, as were patients suffering from diseases, such as Sjogren's syndrome, or with a history of surgery to major salivary glands, or prior head and neck radiotherapy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
plasma nitrate level | one day after nitrate supplementation
  The plasma nitrate level will be determined one day after nitrate supplementation.

SECONDARY OUTCOMES:
quality of life | one day after nitrate supplementation
  The quality of life will be assessed one day after nitrate supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Songlin Wang, Ph.D, Principal Investigator — Professor and Vice President of Capital Medical University
Locations (1):
- Capital Medical University School of Stomatology, Beijing, Beijing Municipality, China